CLINICAL TRIAL: NCT05848193
Title: The Utilization of mHealth Technology to Improve the Treatment and Recovery of Post-concussion Symptoms: A Pilot Randomized Controlled Trial
Brief Title: mHealth Technology in the Treatment of Post-concussion Symptoms
Acronym: PERSIST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Dr. Gihan Perera, Principal Investigator, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16252
Record Dates: First submitted 2023-04-25; First posted 2023-05-08 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Post Concussion Syndrome
MeSH Terms: conditions — Post-Concussion Syndrome | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Patients in the control group will receive standard of care for the treatment of post-concussion symptoms at our Integrated Adult Concussion Clinic
  Interventions: Other: Standard of Care
- mHealth (Experimental): Patients in the intervention group will use MyHeadHealth - an online application to help in the completion of their treatment plan
  Interventions: Other: MyHeadHealth online application

INTERVENTIONS:
Other: MyHeadHealth online application — MyHeadHealth is an online application to be accessed through the patients smartphone. The goal of MyHeadHealth is to improve treatment compliance by providing patients with free and convenient access to resources and activities that align with their treatment plan
  Arms: mHealth
Other: Standard of Care — Patients will receive Standard of Care from our concussion clinic as necessary as per the consultation with the physician
  Arms: Standard of Care

SUMMARY:
Patients with concussion symptoms are asked by their doctors to stretch, exercise, and practice mindfulness daily. Patients can have a hard time sticking to these activities, which can cause patients to feel symptoms for longer than if they stuck to the doctor's suggestions. Many areas of medicine are now using mobile health (mHealth) technology, such as phone applications, to help patients with their treatment plans. No study has looked at the use of phone applications in general population adults with a concussion. This study will look at patient symptoms, quality of life, and satisfaction with care between two groups of patients. Patients will be randomly placed into either the group that gets standard care or the group that will use the smartphone application. The investigators will compare changes in symptoms and quality of life, as well as satisfaction with care, 1 and 3 months after the patient's first visit with their doctor. The investigators hope this study helps to guide the use of mHealth technology in the treatment of post-concussion symptoms.

DETAILED DESCRIPTION:
The proper development of mHealth technology requires the completion of 5 phases as outlined by The Center for eHealth Research and Disease Management. Dr. Perera and his research team have accomplished the first three stages (contextual inquiry, value specification and design); the proposed study will support the completion of phase four (operationalization - the integration of the application into practice) and five (summative evaluation). Using the proposed randomized controlled trial, the investigators will evaluate the use of MyHeadHealth in the rehabilitation of PCS as compared to SOC. While research on the integration of mHealth technology in other health specialties has been beneficial for diagnostic and clinical decision making, behavior change, digital therapeutics and delivering educational content to patients,18 there is a paucity of research in PCS. To properly evaluate the use of mHealth technology in the rehabilitation of PCS, a methodologically robust study directly comparing this new technology to SOC is required. The purpose of this study is to explore the clinical use of MyHeadHealth to treat adult PCS patients. The primary objective of this study is to determine if MyHeadHealth significantly improves patient symptomology when compared to standard of care (SOC). The secondary objective of this study is to understand if MyHeadHealth has a significant effect on treatment compliance, QOL and satisfaction with care as compared to SOC. A sub-group analysis within this study will explore the relationship between self-efficacy and treatment compliance in adult PCS patients.

Patients will be introduced to the study during their consultation with Dr. Perera; if interested, the patient will speak to a research team member and consent to participate. Following consent they will be randomized into their study group and complete the baseline questionnaires. Patients will complete treatment as outlined by their physician. They will be contacted to complete questionnaires at 1 and 3 months following their consultation. Communication will occur via email or mail, depending on how the patient wished to be contacted.

The primary outcome of this study is symptomology. The secondary outcome measures are quality of life, satisfaction with care, self efficacy and treatment compliance.

Data analysis will focus on how the use of MyHeadHealth impacted patient compliance and concomitantly, how that impacted symptoms, quality of life and satisfaction with care. The investigators will also look at the difference in self-efficacy between groups and how that impacted the outcome measures. Within group analyses will also be performed to understand changes within the control and intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Clinician diagnosis of a subconcussive injury or a concussion consistent with the 2017 Berlin Consensus Statement
* Capable of providing consent
* Able to complete study questionnaires
* Fluent in English
* A Glasgow Coma Scale (GCS) score of ≥14
* Has a cellular device that has access to the internet (so they can access MyHeadHealth)

Exclusion Criteria:

* Moderate (GCS 9-13) or Severe (GCS 3-8) Traumatic Brain Injury
* Patients with light sensitivities that prevent looking at devise for longer than 10 minutes
* Patients with a cognitive, physical, or emotional impairment that would prevent them from being able to perform a self-directed program or use the MyHeadHealth app

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Neurobehavioral Symptoms Inventory | Baseline (at consult)
  Measures common symptoms presenting in post-concussion patients- The total scores range from 0-88, with a high score indicative of worse post-concussive symptoms
Neurobehavioral Symptoms Inventory | 1 Month post consult
  Measures common symptoms presenting in post-concussion patients -The total scores range from 0-88, with a high score indicative of worse post-concussive symptoms
Neurobehavioral Symptoms Inventory | 3 Months post consult
  Measures common symptoms presenting in post-concussion patients -The total scores range from 0-88, with a high score indicative of worse post-concussive symptoms

SECONDARY OUTCOMES:
Assessment of Quality-of-Life (AQoL) Scale | Baseline (at consult)
  Measures patient quality of life (physical, emotional and mental) - total score out of 100 - Higher scores represent worsening psychosocial well-being and physical pain
Assessment of Quality-of-Life (AQoL) Scale | 1 month post consult
  Measures patient quality of life (physical, emotional and mental) - total score out of 100 - Higher scores represent worsening psychosocial well-being and physical pain
Assessment of Quality-of-Life (AQoL) Scale | 3 months post consult
  Measures patient quality of life (physical, emotional and mental) - total score out of 100 - Higher scores represent worsening psychosocial well-being and physical pain
Short Assessment of Patient Satisfaction Measure | Baseline (consult)
  Measures Patient Satisfaction with Care - score is totaled with higher scores (maximum of 28) indicating higher levels of satisfaction
Short Assessment of Patient Satisfaction Measure | 1 month post consult
  Measures Patient Satisfaction with Care - score is totaled with higher scores (maximum of 28) indicating higher levels of satisfaction
Short Assessment of Patient Satisfaction Measure | 3 months post consult
  Measures Patient Satisfaction with Care -score is totaled with higher scores (maximum of 28) indicating higher levels of satisfaction
Adapted version of the Morisky Adherence Scale (MMAS-8) | 1 month (post consult)
  Measures patient compliance to treatment plan. Scoring is done by summing questions 1 - 7 and then dividing the score for question 8 by 4 and adding it to the sum of 1-7. High adherence is a score of 8; medium is a score of 6 or 7; low is a score less than 6.
Adapted version of the Morisky Adherence Scale (MMAS-8) | 3 months (post consult)
  Measures patient compliance to treatment plan. Scoring is done by summing questions 1 - 7 and then dividing the score for question 8 by 4 and adding it to the sum of 1-7. High adherence is a score of 8; medium is a score of 6 or 7; low is a score less than 6.
MyHeadHealth tracker | 1 month (post consult)
  Measures patient compliance to treatment plan, headache and sleep quality in patients - randomized to the intervention group - this is not a scale, it is a "bubble sheet" format, where patients fill in a bubble to indicate level of headache, quality of sleep, and compliance to treatment plan
MyHeadHealth tracker | 3 months (post consult)
  Measures patient compliance to treatment plan, headache and sleep quality in patients randomized to the intervention group - this is not a scale, it is a "bubble sheet" format, where patients fill in a bubble to indicate level of headache, quality of sleep, and compliance to treatment plan
Self-Efficacy for Home Exercise Program Scale (SEHEPS) | Baseline (consult)
  Patient Self-Efficacy for Treatment Compliance - a 12-item questionnaire designed to assess perceived self-efficacy for a prescribed home-based exercise plan. For the purposes of this study, the term "exercise plan" was changed to "prescribed treatment plan". Patients answer the questions on a 7-point scale that ranged from 0 (not confident) to 6 (very confident). Total scores ranged from 0 (low self-efficacy) to 72 (high self-efficacy).
Self-Efficacy for Home Exercise Program Scale (SEHEPS) | 1 month (post consult)
  Patient Self-Efficacy for Treatment Compliance - a 12-item questionnaire designed to assess perceived self-efficacy for a prescribed home-based exercise plan. For the purposes of this study, the term "exercise plan" was changed to "prescribed treatment plan". Patients answer the questions on a 7-point scale that ranged from 0 (not confident) to 6 (very confident). Total scores ranged from 0 (low self-efficacy) to 72 (high self-efficacy).
Self-Efficacy for Home Exercise Program Scale (SEHEPS) | 3 months (post consult)
  Patient Self-Efficacy for Treatment Compliance - a 12-item questionnaire designed to assess perceived self-efficacy for a prescribed home-based exercise plan. For the purposes of this study, the term "exercise plan" was changed to "prescribed treatment plan". Patients answer the questions on a 7-point scale that ranged from 0 (not confident) to 6 (very confident). Total scores ranged from 0 (low self-efficacy) to 72 (high self-efficacy).

CONTACTS AND LOCATIONS:
Overall Officials: Gihan Perera, MD, Principal Investigator — McMaster University

IPD SHARING:
Plan to Share IPD: No
We do not plan to make patient data available to other researchers to protect the identity of our patients